CLINICAL TRIAL: NCT00814060
Title: A Single Dose Bioavailability Study of 2 New Tablet Formulations of Neratinib Compared With a Reference Capsule in Healthy Adult Subjects
Brief Title: Study Evaluating TwoTablet Formulations of Neratinib (HKI-272)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-1117
Record Dates: First submitted 2008-12-17; First posted 2008-12-23 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 40-mg tablet
  Interventions: Drug: neratinib
- 2 (Experimental): 240-mg tablet
  Interventions: Drug: neratinib
- 3 (Experimental): 80-mg capsule
  Interventions: Drug: neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
This study will examine the bioavailability (the rate and extent to which the active ingredient or active moiety is absorbed from a drug product and becomes available at the site of action) of two tablet formulations of Neratinib (HKI-272) compared to the capsule formulation.

ELIGIBILITY:
Healthy male and female subjects, ages 18-50.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Blood will be collected to determine the pharmacokinetics of the various formulations of HKI-272 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Tacoma, Washington, United States